CLINICAL TRIAL: NCT05091827
Title: Assessment of the Cardiovascular Risk Profile of Infants Exposed to Pre-eclampsia in Utero
Brief Title: Cardiovascular Risk in Infants Exposed to Pre-eclampsia in Utero
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Walter Sisulu University (Other)
Collaborators: Medical Research Council, South Africa (Other); Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 070/2021
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Offspring of Pre-eclamptic Mothers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pregnant women with pre-eclampsia: Pre-eclamptic pregnant women with singleton uncomplicated ≥ 20 week old pregnancies will be recruited in this group of the study.
- Normotensive pregnant women: Normotensive pregnant women with singleton uncomplicated ≥ 20 week old pregnancies will be recruited in this group of the study
- Offspring of pre-eclamptic women: Both male and female offspring of pre-eclamptic women recruited in this study will be recruited into this study group.
- Offspring of normotensive pregnant women: Both male and female offspring of from normotensive pregnant women recruited in this study will be recruited into this study group.

SUMMARY:
An increasing number of scientific publications show that high blood pressure is being described in younger and younger children of African ancestry. It therefore makes sense to seek for the causes of this raised blood pressure in the in utero events. Recent studies have attributed and increased risk to cardiovascular disease (CVD) risk factors to the gestational environment. Pre-eclampsia (PE) is associated with endothelial dysfunction and oxidative stress in the mother which may influence how the developing foetus interacts with the external environment later on in life. Indeed scientific literature suggests that the foeto-placental vascular endothelial dysfunction may cause epigenetic alteration in the intrauterine environment of the foetus which may be at the origin of chronic diseases in children, thus predisposing them to risk factors of CVD. However, very few studies in women of African ancestry have been carried out to investigate whether or not children born of pre-eclamptic mothers of African ancestry are at risk of developing CVDs. Hence, the aim of this study is to investigate the relationship between pre-eclampsia and cardiovascular risk in children born to pre-eclampsic mothers in a rural South African population. A prospective case-control control design recruiting pre-eclamptic and normotensive pregnant women and their offspring subsequently will be used. CVD risk will be accessed in the pregnant women at 30 weeks of gestation and in the offspring at birth and then six weeks later. The difference in CVD risk between children born to these two groups of women will be assessed and the correlation between maternal and offspring risks for CVDs determined. It is expected that results obtained from this project will provide information on the cardiovascular effect of in utero exposure to PE in a population of African ancestry. This knowledge will advise policy on the management of women with pre-eclampsia with a view of preventing cardiovascular diseases in the offspring. Furthermore, the project will afford the opportunity for scientific research capacity building in students in Walter Sisulu University and foster collaboration between clinical and fundamental researchers.

DETAILED DESCRIPTION:
Study design This will be a prospective case-control study involving babies born to pre-eclamptic (cases) pregnant women as the case and babies born to normotensive mothers (control). The mothers will be recruited at the Nelson Mandela Academic Hospital, Mthatha, Eastern Cape Province of South Africa. This is a tertiary hospital to which all specialist cases are referred from the peripheral hospitals. Even though the prevalence of PE in South Africa is just over 5% nationally, 18% of all obstetric cases consulted in the Nelson Mandela Academic Hospital in Mthatha are PE cases (unpublished data). It will therefore not be a great challenge to recruit the desired number of PE patients over the study period.

Sample size calculation The study done by Amini et al, (2010) showed blood pressure (BP) differences between neonates from normotensive and pre-eclamptic mothers5. The difference in blood systolic BP (SBP) was very high (normotensive: 49.85±5.49 versus pre-eclamptic: 68.2±149). Because the SBP variance and standard deviation were very high in the pre-eclamptic group, we decided to rather use the diastolic blood pressure values (normotensive: 30.17±11.89 versus pre-eclamptic: 42.11±11.49) for sample size calculation. The software - R was used: alpha = 0.01, mean difference = 11.94 and standard = 0.05 respectively were used. The results showed that total sample size is 97 (48 cases and 49 controls). We make the assumption that not all participants would return for the follow-up. Thus we adjusted our sample size by 20% to compensate for possible loses to follow-up. Therefore the total sample will be 97 + (97x20/100) = 117 neonates. However the study will start with the recruitment of 117 pregnant women (58 pre-eclamptic women and 59 normotensive pregnant women who meet the selection criteria).

Ethical approval Ethical approval and permission to carry out the research project has been applied for from Faculty of Health Sciences Research and Ethics Committee (HRSEC) at Walter Sisulu University (WSU). When the project is approved the Provincial and District Departments of Health will be approached for clearance and approval.

Informed consent The purpose of the study will be explained thoroughly to potential participants attending the antenatal clinic in the Nelson Mandela Academic Hospital, Mthatha, Eastern Cape Province. Pregnant women who meet the selection criteria and are willing to participate in the study will be required to sign informed consent forms to participate in the study and to allow their children to participate in the study from birth.

Research Protocol Pregnant women who meet the selection criteria will be recruited between weeks 20-26 of gestation while data will be collected in week 30 of gestation. Participants will be reminded of the hospital visit for data collection in advance to enable them make all necessary preparation to spend some extra time at the hospital.

1. Baseline information: Maternal demographic, obstetric and medical history will be collected from participant using a questionnaire.
2. Anthropometric measurements: Height and weight will be determined as per recommendations of the NHANES, 2009-2010 recommendations24
3. Confirmation of pre-eclampsia status: Hospital files will be used to confirm pre-eclampsia status.
4. Blood pressure measurements: Office blood pressure will be measured as described by Putner et al., (2019)25
5. Flow mediated dilatation. A Mobile Esaote MyLabTM Five portable ultrasound device (Genoa, Italy) with an Esaote Doppler probe (LA523, 12 MHz) connected to computerized software with edge detection technology (Quipu Cardiovascular Suite (CVS)™; Pisa, Italy) will be used. Endothelial function will be measured as described by Strijdom et al (2017)26
6. Gestational ultrasound will be performed to determine placental morphometry, architecture and vascularization. Uterine arteries, umbilical artery and middle cerebral artery will be assessed and uterine artery mean pulsating index determined. Foetal cerebroplacental ratio and anthropometry will be calculated when possible.
7. Measurement of markers of oxidative stress : Fasting blood will be collected for determination of oxidative stress in the maternal environment to which the foetus is exposed.

At birth: The Gestational age at delivery and mode of delivery will be noted. The APGAR score (1-5 minutes), will be determined, weight and height/length of the child will be measured. Cord blood will be collected for determination of titres of CVD risk as indicated below.

1. Markers of endothelial function: Endocan and asymmetric dimethyl arginine (ADMA), markers of endothelial function will be assayed using ELISA kits as per manufacturers' instructions.
2. Markers of oxidative stress: Lipid peroxidation, total antioxidant capacity and 8-hydoxyl-2-deoxyguanine (8-OHdG) will be determined using ELISA kits as per manufacturer's protocols.
3. Lipid profile : Total cholesterol, triglyceride, LDL cholesterol and HDL cholesterol, and oxidised LDL-cholesterol will be measured as per manufacturer's protocol using colorimetric kits as per manufacturers' instructions
4. Insulin Resistance: Fasting glucose, glycated haemoglobin and insulin concentrations will be determined as per manufacturer's methods. The HOMA-IR formula will be used to calculate insulin resistance from fast glucose and insulin as described by Mather et al, 1985)27.
5. Renal function indices: glomerular filtration rate (GFR), creatinine and albumin will be determined using colorimetric kits as per manufacturers' instructions
6. Blood pressure measurements: The oscillometric technique (Dinamap 8100) will be used for BP measurement according to the standard protocol for assessment of BP measurement in newborns by Nwankwo et al. (1997)28.
7. Anthropometric measurements: All measures were done as reported by Meldere et al. (2013) 29.
8. Arterial stiffness will be assessed by measuring Brachio-femoral pulse wave velocity (bfPWV) using an oscillometric device (Vicorder, Skidmore Medical) as reported by Alwan et al., 201530.

ELIGIBILITY:
Inclusion Criteria:

Pre-eclamptic or normotensive pregnant women with singleton uncomplicated ≥ 20 week old pregnancies and their offspring will be recruited for the study.

Exclusion Criteria:

Pregnant women with chronic hypertension, type 2 diabetes, gestational diabetes, renal and cardiovascular diseases or any critical health condition will be excluded from the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pre-eclamptic and normotensive pregnant women and their offspring.
Sampling Method: Probability Sample
Enrollment: 234 (Estimated)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular risk outcomes of children exposed to pre-eclampsia in vitro. | January 2022 to December 2023
  The study will monitor both biochemical and physical risks of cardiovascular risk in exposed children during the second and third trimesters and pregnancy and up to one year after birth.

IPD SHARING:
Plan to Share IPD: No
Data collected from individual participants will be synthesize, analyzed and reported as processed data and not as individual data.

REFERENCES:
- [Background] ACOG Practice Bulletin No. 202 Summary: Gestational Hypertension and Preeclampsia. Obstet Gynecol. 2019 Jan;133(1):1. doi: 10.1097/AOG.0000000000003019. PMID 30575668
- [Background] Bartsch E, Medcalf KE, Park AL, Ray JG; High Risk of Pre-eclampsia Identification Group. Clinical risk factors for pre-eclampsia determined in early pregnancy: systematic review and meta-analysis of large cohort studies. BMJ. 2016 Apr 19;353:i1753. doi: 10.1136/bmj.i1753. PMID 27094586
- [Background] Belay AS, Wudad T. Prevalence and associated factors of pre-eclampsia among pregnant women attending anti-natal care at Mettu Karl referal hospital, Ethiopia: cross-sectional study. Clin Hypertens. 2019 Jul 1;25:14. doi: 10.1186/s40885-019-0120-1. eCollection 2019. PMID 31304042
- [Background] Campos-Canas J, Romo-Palafox I, Albani-Campanario M, Hernandez-Guerrero C. An imbalance in the production of proinflammatory and anti-inflammatory cytokines is observed in whole blood cultures of preeclamptic women in comparison with healthy pregnant women. Hypertens Pregnancy. 2014 May;33(2):236-49. doi: 10.3109/10641955.2013.858744. Epub 2014 Jan 6. PMID 24392828
- [Background] Chambers JC, Fusi L, Malik IS, Haskard DO, De Swiet M, Kooner JS. Association of maternal endothelial dysfunction with preeclampsia. JAMA. 2001 Mar 28;285(12):1607-12. doi: 10.1001/jama.285.12.1607. PMID 11268269
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Background] Craici I, Wagner S, Garovic VD. Preeclampsia and future cardiovascular risk: formal risk factor or failed stress test? Ther Adv Cardiovasc Dis. 2008 Aug;2(4):249-59. doi: 10.1177/1753944708094227. PMID 19124425
- [Background] Friedman SA, Schiff E, Emeis JJ, Dekker GA, Sibai BM. Biochemical corroboration of endothelial involvement in severe preeclampsia. Am J Obstet Gynecol. 1995 Jan;172(1 Pt 1):202-3. doi: 10.1016/0002-9378(95)90113-2. PMID 7847535
- [Background] Leiva A, Pardo F, Ramirez MA, Farias M, Casanello P, Sobrevia L. Fetoplacental vascular endothelial dysfunction as an early phenomenon in the programming of human adult diseases in subjects born from gestational diabetes mellitus or obesity in pregnancy. Exp Diabetes Res. 2011;2011:349286. doi: 10.1155/2011/349286. Epub 2011 Nov 24. PMID 22144986
- [Background] Lowe DT. Nitric oxide dysfunction in the pathophysiology of preeclampsia. Nitric Oxide. 2000 Aug;4(4):441-58. doi: 10.1006/niox.2000.0296. PMID 10944429
- [Background] Maynard SE, Min JY, Merchan J, Lim KH, Li J, Mondal S, Libermann TA, Morgan JP, Sellke FW, Stillman IE, Epstein FH, Sukhatme VP, Karumanchi SA. Excess placental soluble fms-like tyrosine kinase 1 (sFlt1) may contribute to endothelial dysfunction, hypertension, and proteinuria in preeclampsia. J Clin Invest. 2003 Mar;111(5):649-58. doi: 10.1172/JCI17189. PMID 12618519
- [Background] Meeme A, Buga GA, Mammen M, Namugowa A. Endothelial dysfunction and arterial stiffness in pre-eclampsia demonstrated by the EndoPAT method. Cardiovasc J Afr. 2017 Jan/Feb 23;28(1):23-29. doi: 10.5830/CVJA-2016-047. Epub 2016 May 19. PMID 27196639
- [Background] Mol BWJ, Roberts CT, Thangaratinam S, Magee LA, de Groot CJM, Hofmeyr GJ. Pre-eclampsia. Lancet. 2016 Mar 5;387(10022):999-1011. doi: 10.1016/S0140-6736(15)00070-7. Epub 2015 Sep 2. PMID 26342729
- [Background] Nakimuli A, Chazara O, Byamugisha J, Elliott AM, Kaleebu P, Mirembe F, Moffett A. Pregnancy, parturition and preeclampsia in women of African ancestry. Am J Obstet Gynecol. 2014 Jun;210(6):510-520.e1. doi: 10.1016/j.ajog.2013.10.879. Epub 2013 Oct 30. PMID 24184340
- [Background] Noori M, Donald AE, Angelakopoulou A, Hingorani AD, Williams DJ. Prospective study of placental angiogenic factors and maternal vascular function before and after preeclampsia and gestational hypertension. Circulation. 2010 Aug 3;122(5):478-87. doi: 10.1161/CIRCULATIONAHA.109.895458. Epub 2010 Jul 19. PMID 20644016
- [Background] O'Brien M, Baczyk D, Kingdom JC. Endothelial Dysfunction in Severe Preeclampsia is Mediated by Soluble Factors, Rather than Extracellular Vesicles. Sci Rep. 2017 Jul 19;7(1):5887. doi: 10.1038/s41598-017-06178-z. PMID 28725005
- [Background] Muntner P, Shimbo D, Carey RM, Charleston JB, Gaillard T, Misra S, Myers MG, Ogedegbe G, Schwartz JE, Townsend RR, Urbina EM, Viera AJ, White WB, Wright JT Jr. Measurement of Blood Pressure in Humans: A Scientific Statement From the American Heart Association. Hypertension. 2019 May;73(5):e35-e66. doi: 10.1161/HYP.0000000000000087. PMID 30827125
- [Background] Rana S, Lemoine E, Granger JP, Karumanchi SA. Preeclampsia: Pathophysiology, Challenges, and Perspectives. Circ Res. 2019 Mar 29;124(7):1094-1112. doi: 10.1161/CIRCRESAHA.118.313276. PMID 30920918
- [Background] Samanta M, Mondal R, Ray S, Sabui TK, Kundu CK, Hazra A, Chatterjee K, Sarkar D. Blood pressure variation with gestational age and birth weight in Indian newborn. J Trop Pediatr. 2015 Jun;61(3):197-205. doi: 10.1093/tropej/fmv019. Epub 2015 Mar 31. PMID 25833095
- [Background] Schiffrin EL, Flack JM, Ito S, Muntner P, Webb RC. Hypertension and COVID-19. Am J Hypertens. 2020 Apr 29;33(5):373-374. doi: 10.1093/ajh/hpaa057. No abstract available. PMID 32251498
- [Background] Souza JP, Gulmezoglu AM, Vogel J, Carroli G, Lumbiganon P, Qureshi Z, Costa MJ, Fawole B, Mugerwa Y, Nafiou I, Neves I, Wolomby-Molondo JJ, Bang HT, Cheang K, Chuyun K, Jayaratne K, Jayathilaka CA, Mazhar SB, Mori R, Mustafa ML, Pathak LR, Perera D, Rathavy T, Recidoro Z, Roy M, Ruyan P, Shrestha N, Taneepanichsku S, Tien NV, Ganchimeg T, Wehbe M, Yadamsuren B, Yan W, Yunis K, Bataglia V, Cecatti JG, Hernandez-Prado B, Nardin JM, Narvaez A, Ortiz-Panozo E, Perez-Cuevas R, Valladares E, Zavaleta N, Armson A, Crowther C, Hogue C, Lindmark G, Mittal S, Pattinson R, Stanton ME, Campodonico L, Cuesta C, Giordano D, Intarut N, Laopaiboon M, Bahl R, Martines J, Mathai M, Merialdi M, Say L. Moving beyond essential interventions for reduction of maternal mortality (the WHO Multicountry Survey on Maternal and Newborn Health): a cross-sectional study. Lancet. 2013 May 18;381(9879):1747-55. doi: 10.1016/S0140-6736(13)60686-8. PMID 23683641
- [Background] Steegers EA, von Dadelszen P, Duvekot JJ, Pijnenborg R. Pre-eclampsia. Lancet. 2010 Aug 21;376(9741):631-44. doi: 10.1016/S0140-6736(10)60279-6. Epub 2010 Jul 2. PMID 20598363
- [Background] Tessema GA, Tekeste A, Ayele TA. Preeclampsia and associated factors among pregnant women attending antenatal care in Dessie referral hospital, Northeast Ethiopia: a hospital-based study. BMC Pregnancy Childbirth. 2015 Mar 29;15:73. doi: 10.1186/s12884-015-0502-7. PMID 25880924
- [Background] Tooher J, Thornton C, Makris A, Ogle R, Korda A, Hennessy A. All Hypertensive Disorders of Pregnancy Increase the Risk of Future Cardiovascular Disease. Hypertension. 2017 Oct;70(4):798-803. doi: 10.1161/HYPERTENSIONAHA.117.09246. Epub 2017 Sep 11. PMID 28893895
- [Background] Vata PK, Chauhan NM, Nallathambi A, Hussein F. Assessment of prevalence of preeclampsia from Dilla region of Ethiopia. BMC Res Notes. 2015 Dec 24;8:816. doi: 10.1186/s13104-015-1821-5. PMID 26704295
- [Background] Vaughan JE, Walsh SW. Oxidative stress reproduces placental abnormalities of preeclampsia. Hypertens Pregnancy. 2002;21(3):205-23. doi: 10.1081/PRG-120015848. PMID 12517328
- [Background] Weel IC, Baergen RN, Romao-Veiga M, Borges VT, Ribeiro VR, Witkin SS, Bannwart-Castro C, Peracoli JC, De Oliveira L, Peracoli MT. Association between Placental Lesions, Cytokines and Angiogenic Factors in Pregnant Women with Preeclampsia. PLoS One. 2016 Jun 17;11(6):e0157584. doi: 10.1371/journal.pone.0157584. eCollection 2016. PMID 27315098
- [Background] Wu P, Haththotuwa R, Kwok CS, Babu A, Kotronias RA, Rushton C, Zaman A, Fryer AA, Kadam U, Chew-Graham CA, Mamas MA. Preeclampsia and Future Cardiovascular Health: A Systematic Review and Meta-Analysis. Circ Cardiovasc Qual Outcomes. 2017 Feb;10(2):e003497. doi: 10.1161/CIRCOUTCOMES.116.003497. Epub 2017 Feb 22. PMID 28228456